CLINICAL TRIAL: NCT05086211
Title: Comparison of Effects of PNF Techniques and Perturbation Based Balance Training on Risk of Fall and Quality of Life in Elderly Population
Brief Title: PNFand Perturbations Based Exercises on Balance Training in Elder Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Syeda Maria nazir
Record Dates: First submitted 2021-10-19; First posted 2021-10-20 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Balance; Distorted
Keywords: proprioceptive neuromuscular facilitations; pertubation based balance training; elder population
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- proprioceptive neuromuscular facilitation (Experimental): Each session including three PNF techniques:
  Balance training exercises,participants will be treated for 20 minutes with PNF techniques that included;Rhythmic initiation, slow reversal techniques practiced with D1 and D2 pattern in lower limb,repeated contraction and Resisted PNF.The Technique will be performed for 3 days per week in same order on all subjects.
  Interventions: Other: proprioceptive neuromuscular facilitation
- pertubation based balance training (Experimental): Each session will include a 5-10min warm-up,voluntary tasks intended to induce internal perturbations,voluntary tasks combined with external perturbations and a 5-10mins cool down.The technique will be performed for 2 sets of 10 repetitions on all subjects.
  Interventions: Other: pertubation based balance training

INTERVENTIONS:
Other: proprioceptive neuromuscular facilitation — Each session including three proprioceptive neuromuscular facilitation techniques:
  Balance training exercises,participants will be treated for 20 minutes with PNF techniques that included;Rhythmic initiation, slow reversal techniques practiced with D1 and D2 pattern in lower limb,repeated contraction and Resisted PNF.The Technique will be performed for 3 days per week in same order on all subjects.
  Arms: proprioceptive neuromuscular facilitation
Other: pertubation based balance training — Each session will include a 5-10min warm-up,voluntary tasks intended to induce internal perturbations,voluntary tasks combined with external perturbations and a 5-10mins cool down.The technique will be performed for 2 sets of 10 repetitions on all subjects
  Arms: pertubation based balance training

SUMMARY:
To compare the effects of proprioceptive neuromuscular facilitation techniques and perturbation-based balance training on risk of falls and quality of life in elderly population.65 to 85 years old age both male and female participants experienced fall greater than1 time in last 1 year is included in this study.Two groups in this study group A will receive proprioceptive neuromuscular facilitation techniques and group B will receive pertubations based balance training.berg balance scale,time up and go test quality of life scale and Modified John Hopkins Fall Risk Assessment Tool will be used for pre and post assessment.

DETAILED DESCRIPTION:
Balance is very crucial component for living an independent life among older adults and performing their daily life activities independently. Balance control provides foundation to move and perform daily life functions.balance control deteriorates with age, and balance impairment is a major risk of fall among older adults. Fall may result in severe injuries, fracture, causing severe longstanding pain, low quality of life, disability or death. In older adults, falls most commonly result in many co-morbidities and mortality. The proprioceptive Neuromuscular Facilitation is greatly used technique as an intervention for neuromuscular dysfunction. By applying PNF technique, therapist can improve movement re-education.this technique help in improving muscle strengthening and stabilization. PNF technique uses reflexes of nervous system that help to relax a muscle.proprioceptive neuromuscular facilitation (PNF) promotes strengthening, motor learning and restoration of motor control in elderly individuals despite of neuromuscular and deficits.The Perturbation-based balance training comprises of some unpredictable, multi-directional dynamic-platform perturbations to elicit stepping and grasping reactions. The extent of perturbations is gradually improved over the period of program. The perturbation-based balance training program can help to improve or reverse impairments associated with older age in balance-recovery reactions. This program will greatly help in preventing falls, which may lead to improved health, enhanced mobility, more independence and high quality of life. Increased frequency of collisions are shown by older adults in swing phase and stance leg. Moreover, step length is also reduced and the frequency of multiple-step responses is increased. Older individuals rely more upon arm reactions to recover balance but the speed tends to decrease while initiation and execution of grasping reaction. And all reactions mentioned above are associated with increased risk of falling. The perturbation-based training program promote effective change in support program reactions that may help to reduce risk of falls and this training program should be part of fall prevention program and thus helping in improved quality of life

ELIGIBILITY:
Inclusion Criteria:

* 65 years - 85 years of age
* Gender: Both Male and Female
* Participants experienced fall >1 time in last 1 year.
* Patients should stand independently without upper limb support for >30s.
* Participants should tolerate at least 10 postural perturbations.

Exclusion Criteria:

* Participants with body weight > 100kgs.
* Participants with lower extremity amputation.
* Severe osteoporosis
* Having recent illness, surgery, cognitive impairment or another neurological deficit.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-06-26 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-08-15 (Actual)

PRIMARY OUTCOMES:
berg balance scale | week 6
  Berg Balance Scale is the gold standard scale for assessment of Static and Dynamic Balance of a person. It is widely used in clinical settings. It consists of 14 balance related tasks. If a person performs the task independently it means a score of 4 and if a person is unable to do a task then a score of 0 is given. The sum of all the scores at the end will give us a final measure. It is a valid and reliable tool.

SECONDARY OUTCOMES:
Time up and Go Test | week 6
  it is a test used to assess the mobility of an individual. It requires the assessment of both static and dynamic balance. It is a reliable and valid tool.
Quality of life Scale | week 6
  It is a 16-item scale used to assess the quality of life. It is internally consistent (a=0.82 to 0.92 with a test-retest reliability of r=0.78 to 0.84)
Modified John Hopkins Fall Risk Assessment Tool | week 6
  This is a simple tool used for assessment of risk of fall in older adults. It is a multifactor tool with promising sensitivity and specificity. It consists of 7 components. Its Inter-rater reliability is 85.7%

CONTACTS AND LOCATIONS:
Overall Officials: Sania Aziz, MSNMPT, Principal Investigator — Riphah International University
Locations (1):
- Muzzaffar Khan Surgical Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Halvarsson A, Dohrn IM, Stahle A. Taking balance training for older adults one step further: the rationale for and a description of a proven balance training programme. Clin Rehabil. 2015 May;29(5):417-25. doi: 10.1177/0269215514546770. Epub 2014 Sep 8. PMID 25200877
- [Background] Mansfield A, Peters AL, Liu BA, Maki BE. A perturbation-based balance training program for older adults: study protocol for a randomised controlled trial. BMC Geriatr. 2007 May 31;7:12. doi: 10.1186/1471-2318-7-12. PMID 17540020
- [Background] Guirguis-Blake JM, Michael YL, Perdue LA, Coppola EL, Beil TL. Interventions to Prevent Falls in Older Adults: Updated Evidence Report and Systematic Review for the US Preventive Services Task Force. JAMA. 2018 Apr 24;319(16):1705-1716. doi: 10.1001/jama.2017.21962. PMID 29710140
- [Background] Beling J, Roller M. Multifactorial intervention with balance training as a core component among fall-prone older adults. J Geriatr Phys Ther. 2009;32(3):125-33. doi: 10.1519/00139143-200932030-00008. PMID 20128337
- [Background] Dunsky A. The Effect of Balance and Coordination Exercises on Quality of Life in Older Adults: A Mini-Review. Front Aging Neurosci. 2019 Nov 15;11:318. doi: 10.3389/fnagi.2019.00318. eCollection 2019. PMID 31803048
- [Background] Heydarnejad S, Dehkordi AH. The effect of an exercise program on the health-quality of life in older adults. A randomized controlled trial. Dan Med Bull. 2010 Jan;57(1):A4113. PMID 20175947
- [Background] You H, Zhang H, Liu J, Han T, Zhang M, Zhao W, Jiang S. Effect of balance training with Pro-kin System on balance in patients with white matter lesions. Medicine (Baltimore). 2017 Dec;96(51):e9057. doi: 10.1097/MD.0000000000009057. PMID 29390433
- [Background] Godi M, Franchignoni F, Caligari M, Giordano A, Turcato AM, Nardone A. Comparison of reliability, validity, and responsiveness of the mini-BESTest and Berg Balance Scale in patients with balance disorders. Phys Ther. 2013 Feb;93(2):158-67. doi: 10.2522/ptj.20120171. Epub 2012 Sep 27. PMID 23023812
- [Background] Hnizdo S, Archuleta RA, Taylor B, Kim SC. Validity and reliability of the modified John Hopkins Fall Risk Assessment Tool for elderly patients in home health care. Geriatr Nurs. 2013 Sep-Oct;34(5):423-7. doi: 10.1016/j.gerinurse.2013.05.011. Epub 2013 Jun 29. PMID 23816376
- [Background] Seo KC, Kim HA. The effects of ramp gait exercise with PNF on stroke patients' dynamic balance. J Phys Ther Sci. 2015 Jun;27(6):1747-9. doi: 10.1589/jpts.27.1747. Epub 2015 Jun 30. PMID 26180312